CLINICAL TRIAL: NCT06401473
Title: Closing the Gate: Investigating a No-Cost, Noninvasive, Patient-Driven Approach to Pain Reduction for Trigger Finger Injections
Brief Title: Using the Gate Control Theory of Pain to Decrease Pain During Trigger Finger Corticosteroid Injections
Acronym: TFGCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Canyon University (Other)
Responsible Party: Principal Investigator, Aidan Crislip, Principal Investigator, Grand Canyon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2023-5842
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Trigger Finger; Pain
Keywords: Gate Control Theory of Pain; Injection
MeSH Terms: conditions — Trigger Finger Disorder; Pain

STUDY DESIGN:
Intervention Model Description: Random assignment into one of three parallel groups: control, distraction, or experimental
Who Masked: Participant
Masking Description: Patients remained blinded to their assigned intervention until after all study procedures were complete.
  Injecting provider was technically blinded but was functionally unblinded at the time of the injection itself due to the visible and audible differences between each group throughout the course of the injection.
  Outcome assessor was blinded while instructing patients how to denote their pain level after the procedure, but was unblinded at the time of the injection. No input was given by the outcome assessor after they were unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients received no intervention during cortisone injection.
- Distraction (Sham Comparator): Patients were instructed on a sham motor distraction task on the contralateral upper limb and performed this task during cortisone injection.
  Interventions: Behavioral: Motor Distraction Task
- Experimental (Experimental): Patients were instructed on the experimental task, involving scratching the upper limb ipsilateral to the site of the injection, and they performed this task during cortisone injection.
  Interventions: Behavioral: Ipsilateral Scratch Task

INTERVENTIONS:
Behavioral: Ipsilateral Scratch Task — Patients scratch the skin within the relevant cervical dermatome, ipsilateral to the injection site
  Arms: Experimental
Behavioral: Motor Distraction Task — Patients scratch the skin of the shoulder/neck contralateral to the injection site
  Arms: Distraction

SUMMARY:
The goal of this clinical trial is to investigate a new noninvasive technique that patients may use to help reduce the pain that they experience during cortisone injections for trigger fingers. It will also help provide information that may help support the gate control theory of pain as a framework for understanding and managing acute pain.The main questions it aims to answer are:

Can a physical stimulus near the site of cortisone injection reduce the pain experienced by the patient during the injection? Does the physical stimulation or the cognitive distraction contribute more to pain relief?

Researchers will compare a physical stimulus near the injection site to a placebo (a similar task that theoretically should not reduce the experience of pain) to see if physical stimuli work to improve pain during injections.

Participants will:

Estimate how much pain they expect to experience during a cortisone injection Receive a cortisone injection for a trigger finger while performing one of three possible actions (control, placebo task, or the investigated physical stimulus near the injection site) Express how much pain they actually experienced during the injection

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age.
* Have been diagnosed with one or more "trigger fingers" of the index, middle, ring, or small fingers.
* Have decided to try a cortisone injection for one or more trigger fingers today as advised by your physician.
* Are able to read and understand these study procedures.

Exclusion Criteria:

* Are severely visually impaired.
* Have a history of spinal cord injury.
* Have taken opioid pain medications in the last 28 days.
* Are currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Score | Immediately after injection (within 10 seconds)
  Patients denote the pain they experienced during the injection based on a standard 100-mm Visual Analog Scale. Scores range from 0-100, with lower scores indicating less pain. A score of 0 indicates no pain at all, while a score of 100 indicates the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Aidan Crislip, BS, Principal Investigator — Grand Canyon University
Locations (1):
- OrthoArizona, Gilbert, Arizona, United States

IPD SHARING:
Plan to Share IPD: No